CLINICAL TRIAL: NCT03510104
Title: A Phase I Dose Escalation Study of the Safety, Pharmacokinetics and Pharmacodynamics of MRX-2843 in Adult Subjects With Relapsed/Refractory Advanced and/or Metastatic Solid Tumors
Brief Title: Pharmacokinetic and Safety Study of MRX-2843 in Adults With Relapsed/Refractory Advanced and/or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meryx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2843-1001
Record Dates: First submitted 2018-04-16; First posted 2018-04-27 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Advanced Cancer; Metastatic Cancer; Neoplasms; Neoplasm Metastasis; Neoplastic Processes; Pathologic Processes
Keywords: MerTK
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Neoplastic Processes; Pathologic Processes | interventions — MRX-2843

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MRX-2843 (Experimental): MRX-2843: Dose Escalation Successive dose escalation cohorts to determine MTD
  Interventions: Drug: MRX-2843

INTERVENTIONS:
Drug: MRX-2843 — MRX-2843 capsules

SUMMARY:
This first-in-human open-label, dose escalation study is designed to evaluate the safety, tolerability, and PK of MRX-2843 in subjects with relapsed/refractory advanced and/or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age.
* Histologically or cytologically confirmed, measurable (defined as those that could be accurately measured in a least 1 dimension with a longest diameter ≥20 mm using conventional techniques or ≥10 mm with spiral computed tomography scan) or evaluable solid malignancy (with the exception of primary central nervous system [CNS] tumors) per RECIST 1.1. Scans performed within 1 month of starting study drug will be accepted.
* Received at least one systemic therapy for advanced disease, with no further approved treatment options that provide proven clinical benefit.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Females of childbearing potential who are sexually active with a nonsterilized male partner agree to use 2 methods of effective contraception from screening, and agree to continue using such precautions for 90 days after the final dose of study drug; cessation of birth control after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control.
* Nonsterilized males who are sexually active with a female of childbearing potential must agree to use an acceptable method of effective contraception from Day 1 and for 90 days after the final dose of study drug.
* Female subjects of childbearing potential must be nonpregnant, nonlactating, and have a negative pregnancy test result at Screening and Day 1 of Cycles 1-6.
* Able to provide written, informed consent before initiation of any study related procedures, and is able, in the opinion of the Investigator, to comply with all the requirements of the study.
* Able to swallow oral medication.
* Subject has the following laboratory values at Screening:

  1. Absolute neutrophil count ≥1500/mm3
  2. Platelet count ≥100,000/mm3
  3. Hemoglobin ≥9.0 g/dL (must be >2 weeks post-red blood cell transfusion)
  4. Bilirubin ≤1.5x the upper limit of normal (ULN). For subjects with documented Gilbert's disease, bilirubin ≤3.0 mg/dL. For subjects with documented liver metastases, bilirubin ≤ 2.5x ULN.
  5. Serum creatinine ≤1.5x the ULN or creatinine clearance (CrCl) ≥50 mL/min.
  6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3x the ULN (≤5x the ULN for subjects with liver metastases)

Exclusion Criteria:

* Subject has an abnormal electrocardiogram (ECG) that, in the Investigator's opinion, is clinically significant and would preclude study participation.
* Subject has QT interval corrected (QTc) >480 ms (both males and females) at Screening (repeat values may be obtained during the period between Screening and admission to the study site).
* Subject has any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion of the study drug, or any other condition that may place the subject at risk for such interference (for example, short bowel syndrome or inflammatory bowel disease).
* Subject has a history of Type 1 Diabetes (T1D) or is considered at high risk for T1D, where high risk is defined as

  1. Subject has 1 first-degree relative (FDR; defined as parents, offspring or siblings) with T1D AND A1C value > 6.5% or
  2. Subject has 2+FDR with T1D
* Subject has uncontrolled hypertension, defined as a blood pressure reading >160/100 mmHg, despite maximum antihypertensive therapy.
* Subject has received:

  1. Radionuclide treatment within 6 weeks of the first dose of study drug in this study
  2. Local palliative radiation therapy (XRT) (small port) ≤2 weeks before first dose of study drug
  3. Treatment with therapeutic doses of metaiodobenzylguanidine (MIBG) ≤6 weeks before first dose of study drug
  4. Prior total body irradiation, total craniospinal XRT, or ≥50% radiation of pelvis within 6 months of receiving first dose of study drug
  5. Treatment with a monoclonal antibody within 28 days or 5 half-lives, whichever is shorter, from treatment with first dose of study drug
  6. Therapy with a growth factor within 7 days of starting study drug
  7. Chemotherapy within 3 weeks of starting study drug (6 weeks if prior nitrosourea)
  8. Subjects receiving systemic (oral or parenteral) corticosteroid therapy within 7 days of first dose of study drug or a requirement for chronic systemic immunosuppressive therapy for any reason. Topical or inhaled steroids are allowed.
* Subject has not fully recovered to baseline or National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) ≤ Grade 1 from toxicity due to all prior therapies, except alopecia and other non-clinically significant AEs.
* Subject has any history of human immunodeficiency virus (HIV) or immunodeficiency at Screening.
* Subject has a diagnosis of chronic active hepatitis B or C.
* Subject has uncontrolled intercurrent illness including, but not limited to ongoing or active bacterial, fungal, or viral infection requiring intravenous therapy (not prophylaxis) at the time of study enrollment, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subject has a history of a major adverse cardiac event, including cerebrovascular accident or myocardial infarction within the prior 6 months, or uncontrolled congestive heart failure (New York Heart Association class 3 or 4) at Screening.
* Subject has active, suspected, or previously documented autoimmune disease, defined as requiring systemic treatment.
* Subject has known or suspected history of retinitis pigmentosa or known or suspected familial history of retinitis pigmentosa.
* Subject has prothrombin time/International Normalized Ratio or partial thromboplastin time test results at screening ≥1.5 x ULN.
* Subject requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin-related agents, thrombin or FXa inhibitors, or antiplatelet agents (eg, clopidogrel). Low-dose aspirin (≤81 mg/day), low-dose warfarin (≤1 mg/day), and prophylactic low molecular weight heparin are permitted.
* Subject had surgery (excluding line insertions) within 1 month of the first dose of study drug or has lingering wound complications.
* Subject is unable or unwilling to abide by the study protocol or cooperate fully with the Investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with Dose Limiting Toxicities (DLTs) | Baseline to the end of Cycle 1 (up to 28 days)
Percentage of subjects with Adverse Events (AEs) and Serious Adverse Events (SAEs) graded per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5 | Baseline up to 14 days after last dose of study treatment (up to approximately 12 months)

SECONDARY OUTCOMES:
Determine Maximum Tolerated Dose (MTD) in mg of MRX-2843 | Baseline to end of Cycle 1 (up to 28 days)
AUC0-t: area under the concentration-time curve from time 0 to the time of the last quantifiable concentration (t) | Day 1 and Day 16 of Cycle 1
AUC0-inf: area under the concentration-time curve from time 0 to infinity | Day 1 and Day 16 of Cycle 1
AUC0-τ: area under the concentration-time curve from time 0 to tau, where tau is the dosing interval | Day 1 and Day 16 of Cycle 1
Cmax: maximum observed plasma concentration | Day 1 and Day 16 of Cycle 1
Tmax: time to reach maximum observed plasma concentration | Day 1 and Day 16 of Cycle 1
λz: terminal phase elimination rate constant | Day 1 and Day 16 of Cycle 1
t1/2: apparent terminal elimination half-life | Day 1 and Day 16 of Cycle 1
CL/F: apparent total body clearance | Day 1 and Day 16 of Cycle 1
Vz/F: apparent volume of distribution of the terminal phase | Day 1 and Day 16 of Cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Donald Harvey, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No